CLINICAL TRIAL: NCT00391157
Title: VELCADEXA: A National, Multi-Center, Open-Label Study of Pretransplant Induction With Alternating VELCADE and Dexamethasone (VEL/Dex) in Younger (< 65 Yrs) Untreated Multiple Myeloma Patients.
Brief Title: VELCADEXA: Velcade and Dexamethasone in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-000186-19; VELCADEXA
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Multiple Myeloma
Keywords: Múltiple Myeloma; Transplant; Patients <65 years.
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone

INTERVENTIONS:
Drug: Velcade/Dexamethasone — Velcade 1,3 mg/m2 on days 1, 4, 8 and 11

SUMMARY:
The primary efficacy objective of this study is to study the efficacy in terms of response rate to alternating bortezomib/dexamethasone regimen

DETAILED DESCRIPTION:
Multiple Myeloma is a plasma cell disorder characterized by an uncontrolled proliferation of bone marrow plasma cells leading to skeletal destruction with bone pain, anemia, renal failure, hypercalcemia, recurrent bacterial infections and extramedullary plasmacytomas. It accounts for 1% of all malignancies and slightly more than 10% of hematologic malignancies, with an annual incidence of about four per 100.000. Although this disease is incurable with a median survival of about 3 years, remarkable treatment advances have been recently made, including high-dose therapy followed by stem cell rescue and, particularly, the introduction of novel promising agents with new mechanisms of action.

Data from pre-clinical and clinical studies conducted to date support the continued development of VELCADE for the treatment of Multiple Myeloma. Standard chemotherapy remains as the gold standard for induction before HDT/SCT treatment in younger multiple myeloma patients (<65 years). Since VELCADE has a mechanism of action different from chemotherapy and dexamethasone and is considered to be efficacious in Multiple Myeloma, its introduction in induction regimens may contribute to increase the response rate and eventually survival of these patients that represent half of myeloma population.

Since VBMCP/VBAD is considered to be the gold standard for Multiple Myeloma patients <65 years as induction regimen prior HDT/SCT, the results of VEL/DEX will be compared with those obtained in 100 patients treated with VBMCP/VBAD chemotherapy in our last GEM protocol (Spanish Myeloma Group) for patients <65 years (closed in Dec 2004

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Age over 18 and under 65 years old.
* Patient recently diagnosed with symptomatic Multiple Myeloma based on standard criteria and that has not received any previous chemotherapy treatment for Multiple Myeloma.
* Patient has measurable disease, defined as follows:

For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value and, where applicable, urine light-chain excretion of ≥ 200 mg/24 hours.

For poor or non-secretory multiple myeloma, measurable disease is defined by the presence of soft tissue (not bone) plasmacytomas as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan). In patients with oligosecretory multiple myeloma, the serum and/or urine M-protein measurements are very low and difficult to follow for response assessment. In patients with non-secretory multiple myeloma, there is no M-protein in serum or urine by immunofixation.

* Patient has a ECOG performance status < 2.
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values within 14 days before Baseline visit (Day 1 of Cycle 1, before study drug administration):

Platelet count ≥ 50x109/L, hemoglobin ≥ 8 g/dl and absolute neutrophil count (ANC) ≥ 1.0x109/L; Corrected serum calcium <14mg/dl. Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal. Alanine transaminase (ALT): ): ≤ 2.5 x the upper limit of normal. Total bilirubin: ≤1.5 x the upper limit of normal. Serum creatinine value ≤ 2mg/dl

Exclusion Criteria:

* Patient previously received treatment with VELCADE.
* Patient previously received treatment for Multiple Myeloma
* Patient had major surgery within 4 weeks before enrollment.
* Patient has a platelet count < 50x 109/L within 14 days before enrollment.
* Patient has an absolute neutrophil count < 1.0 x 109/L within 14 days before enrollment.
* Patient has < Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Patient has received other investigational drugs within 14 days before enrollment.
* Patient is known to be seropositive for the human immunodeficiency virus (HIV), Hepatitis B surface antigen-positive or active hepatitis C infection.
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.
* Pregnancy, breast-feeding or fertile women who are not going to use a medical effective contraceptive method during the trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months

SECONDARY OUTCOMES:
Compare the efficacy of velcade and dexamethasone with chemotherapy combination VBMCP/VBAD | 1 year
Evaluate the quality of progenitors cells after treatment with Velcade and dexamethasone | 6 months
Compare the complete response rate after high dose therapy in patients treated with velcade and dexamethasone or VBMCP/VBAD | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bladé Joan, Dr, Study Chair — Hospital Clinic of Barcelona
Locations (10):
- Spain (10):
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona, Barcelona
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital La Fe, Valencia, Valencia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital General de Segovia, Segovia

REFERENCES:
- [Background] Longo D. Plasma cell disorders. In: Fauce A, et al. Ed. Harrison's Principles of Internal Medicine. 14th Ed. New York, New York: Mc Graw-Hill; 1998: 712-718.
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] Raje N, Anderson K. Thalidomide--a revival story. N Engl J Med. 1999 Nov 18;341(21):1606-9. doi: 10.1056/NEJM199911183412110. No abstract available. PMID 10564693
- [Background] Oken MM. Management of Myeloma: Current and Future Approaches. Cancer Control. 1998 May;5(3):218-225. doi: 10.1177/107327489800500302. PMID 10761055
- [Background] Westin J. Conventional chemotherapy in multiple myeloma. Pathol Biol (Paris). 1999 Feb;47(2):169-71. PMID 10192883
- [Background] Huang YW, Hamilton A, Arnuk OJ, Chaftari P, Chemaly R. Current drug therapy for multiple myeloma. Drugs. 1999 Apr;57(4):485-506. doi: 10.2165/00003495-199957040-00004. PMID 10235689
- [Background] Smith ML, Newland AC. Treatment of myeloma. QJM. 1999 Jan;92(1):11-4. doi: 10.1093/qjmed/92.1.11. PMID 10209667
- [Background] Bataille R, Harousseau JL. Multiple myeloma. N Engl J Med. 1997 Jun 5;336(23):1657-64. doi: 10.1056/NEJM199706053362307. No abstract available. PMID 9171069
- [Background] Alexanian R, Dimopoulos M. The treatment of multiple myeloma. N Engl J Med. 1994 Feb 17;330(7):484-9. doi: 10.1056/NEJM199402173300709. No abstract available. PMID 8289856
- [Background] Gregory WM, Richards MA, Malpas JS. Combination chemotherapy versus melphalan and prednisolone in the treatment of multiple myeloma: an overview of published trials. J Clin Oncol. 1992 Feb;10(2):334-42. doi: 10.1200/JCO.1992.10.2.334. PMID 1531068
- [Background] Case DC Jr, Lee DJ 3rd, Clarkson BD. Improved survival times in multiple myeloma treated with melphalan, prednisone, cyclophosphamide, vincristine and BCNU: M-2 protocol. Am J Med. 1977 Dec;63(6):897-903. doi: 10.1016/0002-9343(77)90543-5. No abstract available. PMID 605911
- [Background] Alexanian R, Barlogie B, Tucker S. VAD-based regimens as primary treatment for multiple myeloma. Am J Hematol. 1990 Feb;33(2):86-9. doi: 10.1002/ajh.2830330203. PMID 2301376
- [Background] Alexanian R, Dimopoulos MA, Delasalle K, Barlogie B. Primary dexamethasone treatment of multiple myeloma. Blood. 1992 Aug 15;80(4):887-90. PMID 1498331
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Alexanian R, Weber D, Giralt S, Dimopoulos M, Delasalle K, Smith T, Champlin R. Impact of complete remission with intensive therapy in patients with responsive multiple myeloma. Bone Marrow Transplant. 2001 May;27(10):1037-43. doi: 10.1038/sj.bmt.1703035. PMID 11438818
- [Background] Nadal E, Gine E, Blade J, Esteve J, Rosinol L, Fernandez-Aviles F, Marin P, Martinez C, Rovira M, Urbano-Ispizua A, Carreras E, Montserrat E. High-dose therapy/autologous stem cell transplantation in patients with chemosensitive multiple myeloma: predictors of complete remission. Bone Marrow Transplant. 2004 Jan;33(1):61-4. doi: 10.1038/sj.bmt.1704313. PMID 14704657
- [Background] Driscoll J. The role of the proteasome in cellular protein degradation. Histol Histopathol. 1994 Jan;9(1):197-202. PMID 8003815
- [Background] Richter-Ruoff B, Wolf DH. Proteasome and cell cycle. Evidence for a regulatory role of the protease on mitotic cyclins in yeast. FEBS Lett. 1993 Dec 20;336(1):34-6. doi: 10.1016/0014-5793(93)81603-w. PMID 8262212
- [Background] Goldberg AL, Stein R, Adams J. New insights into proteasome function: from archaebacteria to drug development. Chem Biol. 1995 Aug;2(8):503-8. doi: 10.1016/1074-5521(95)90182-5. PMID 9383453
- [Background] Hideshima T, Richardson P, Chauhan D, Palombella VJ, Elliott PJ, Adams J, Anderson KC. The proteasome inhibitor PS-341 inhibits growth, induces apoptosis, and overcomes drug resistance in human multiple myeloma cells. Cancer Res. 2001 Apr 1;61(7):3071-6. PMID 11306489
- [Background] Sherr CJ. Cancer cell cycles. Science. 1996 Dec 6;274(5293):1672-7. doi: 10.1126/science.274.5293.1672. PMID 8939849
- [Background] Koepp DM, Harper JW, Elledge SJ. How the cyclin became a cyclin: regulated proteolysis in the cell cycle. Cell. 1999 May 14;97(4):431-4. doi: 10.1016/s0092-8674(00)80753-9. No abstract available. PMID 10338207
- [Background] Read MA, Neish AS, Luscinskas FW, Palombella VJ, Maniatis T, Collins T. The proteasome pathway is required for cytokine-induced endothelial-leukocyte adhesion molecule expression. Immunity. 1995 May;2(5):493-506. doi: 10.1016/1074-7613(95)90030-6. PMID 7538441
- [Background] Palombella VJ, Rando OJ, Goldberg AL, Maniatis T. The ubiquitin-proteasome pathway is required for processing the NF-kappa B1 precursor protein and the activation of NF-kappa B. Cell. 1994 Sep 9;78(5):773-85. doi: 10.1016/s0092-8674(94)90482-0. PMID 8087845
- [Background] Zetter BR. Adhesion molecules in tumor metastasis. Semin Cancer Biol. 1993 Aug;4(4):219-29. PMID 8400144
- [Background] Beg AA, Baltimore D. An essential role for NF-kappaB in preventing TNF-alpha-induced cell death. Science. 1996 Nov 1;274(5288):782-4. doi: 10.1126/science.274.5288.782. PMID 8864118
- [Background] Baldwin AS. Control of oncogenesis and cancer therapy resistance by the transcription factor NF-kappaB. J Clin Invest. 2001 Feb;107(3):241-6. doi: 10.1172/JCI11991. No abstract available. PMID 11160144
- [Background] McConkey DJ, Pettaway C, Elliott P, et al. The proteasome as a new drug target in metastatic prostate cancer. ATMDACC 7th Annual Genitourinary Oncology Conference, 1998.
- [Background] Adams J, Palombella VJ, Sausville EA, Johnson J, Destree A, Lazarus DD, Maas J, Pien CS, Prakash S, Elliott PJ. Proteasome inhibitors: a novel class of potent and effective antitumor agents. Cancer Res. 1999 Jun 1;59(11):2615-22. PMID 10363983
- [Background] Millenium Pharmaceuticals, Inc. (PS-341) Investigator's Brochure, Version 5.0, 2001
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- See also: Spanish association of Haematology — http://www.aehh.org